CLINICAL TRIAL: NCT01294475
Title: Preventing Child Maltreatment Through A Cellular-Phone Technology-Based Parenting Program
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-5054
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Child Maltreatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cell Phone Enhanced Parent Training (Experimental): Cell phones will be provided to mothers participating in Planned Activities Training.
  Interventions: Behavioral: Planned Activities Training

INTERVENTIONS:
Behavioral: Planned Activities Training — Mothers will be provided a parenting intervention, Planned Activities Training (PAT). Some of the mothers will receive the PAT intervention enhanced with a cell phone.

SUMMARY:
The goal of this project is to examine the effects of the use of cellular-phone technology in conjunction with a parenting program entitled "Planned Activities Training (PAT)" on participant enrollment, engagement, and motivation for the PAT intervention, as well as on parent and child outcomes.

DETAILED DESCRIPTION:
The current project will employ a 3-group experimental design with random assignment of parents to one of three groups: Planned Activities Training as usual (PAT); Cellular Phone Enhanced PAT (CPAT), or a no-intervention control group. Two cohorts of high-risk mother-child dyads (low education or mother adolescent at time of birth) will be recruited. In years 1 and 2, the first cohort of participants will be recruited in Kansas City, MO and South Bend, IN from an ongoing longitudinal descriptive study of child neglect, which has tracked risk and protective factors since the child's birth (n=180). During years 3 and 4, a second cohort of matched high risk mothers (operationally defined the same as for cohort 1) will be recruited from Head Start programs within the same two communities (n=180). Families in both cohorts will be enrolled when the first family child is between the ages of 4 and 6 years.

Participants assigned to the intervention groups will receive intervention services in the home setting and will be assessed prior to the intervention, as well as at 1-, 6-, and 12- month post-intervention time points. The control group participants will complete assessments at similar time points to the intervention groups. Several outcomes will be examined in order to measure intervention effects, including child maltreatment risk and occurrences, parent behaviors, and child behaviors. These outcomes will be collected utilizing a multi-method approach that will involve parent interview, parent-report and self-report measures, mother-child observation, and review of local CPS system records. For those parents participating in an intervention group, data will also be collected on maternal engagement, retention, fidelity, and dosage with regard to the intervention. Lastly, program and participant costs will be examined to determine the cost-effectiveness of including a technological component with this existing parenting program. It is expected that the knowledge generated through this study will aid in the improvement of parenting interventions targeting the prevention of child maltreatment.

ELIGIBILITY:
Inclusion:

* Women between the ages of 15-18 at the time of their first child's birth OR between the ages of 22-35 years at the time of their first child's birth, with no formal education beyond high school or GED
* Mothers' oldest biological child should be between 4 and 6 years
* Families anticipate living in the 50 mile vicinity of Kansas City or South Bend for the next 18 months
* Primary caregiver should be functionally literate.
* Must speak English or Spanish fluently.

Exclusion:

* Mother has a major medical illness that could interfere with her ability to participate in a 2-year project
* Mother currently lives in a treatment program or rehab center
* Mother has a serious mental illness
* Mother lives in a group home or correctional program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2007-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Child Maltreatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Judy Carta, Ph.D., Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

REFERENCES:
- [Derived] Carta JJ, Lefever JB, Bigelow K, Borkowski J, Warren SF. Randomized trial of a cellular phone-enhanced home visitation parenting intervention. Pediatrics. 2013 Nov;132 Suppl 2(Suppl 2):S167-73. doi: 10.1542/peds.2013-1021Q. PMID 24187120